CLINICAL TRIAL: NCT04999670
Title: Post-operative Pain in Patients Undergoing Caesarean Section: Randomised Trial Evaluating Three Methods of Fascial Closure
Brief Title: Fascial Closure and Post-caesarean Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Richard Pittini, Obstetrician and Gynaecologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FAS-101
Record Dates: First submitted 2020-12-22; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy Related; Cesarean Section; Post-operative Pain; Fascial Closure; Surgical Technique
Keywords: Pregnancy-Related; Cesarean Section; Post-operative Pain; Fascial Closure; Surgical Technique
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomised into one of three groups based upon the method of fascial closure prior to their caesarean section.
Who Masked: Participant, Investigator
Masking Description: Participants will not be made aware which method of fascial closure group they will be in, and investigators will also be blinded to the method of fascial closure as they approach participants to fill in their follow-up questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single suture, knot above fascia (Active Comparator): Fascia sutured with #1 polysorb braided absorbable suture, with the knot being superficial to the fascia, starting at the left angle of the fascial incision and closed in a continuous fashion. The contralateral angle is grasped with a kocher clamp and the suture is then tied behind the angle ensuring adequate closure.
  Interventions: Procedure: Fascial closure method during caesarean section via pfannenstiel incision.
- Two sutures, knot above fascia (Active Comparator): Fascia sutured using #1 polysorb braided absorbable suture with a superficial knot, starting at the left angle and closed in a continuous fashion until the suture is above the right rectus abdominis muscle belly. A second #1 polysorb braided absorbable suture is tied behind the right angle with a superficial knot and run across in a continuous fashion to meet the opposing suture which are then tied together.
  Interventions: Procedure: Fascial closure method during caesarean section via pfannenstiel incision.
- Two sutures, buried knots below fascia (Active Comparator): Fascia sutured using #1 polysorb braided absorbable suture with a buried knot below the fascia starting at the left angle and closed in a continuous fashion until the suture overlies the right rectus abdominis muscle belly. A second #1 polysorb braided absorbable suture is then tied behind the right angle with a buried knot below the fascia and run across in a continuous fashion to meet the opposing suture which are then tied together.
  Interventions: Procedure: Fascial closure method during caesarean section via pfannenstiel incision.

INTERVENTIONS:
Procedure: Fascial closure method during caesarean section via pfannenstiel incision. — Comparison of three different methods of fascial closure.

SUMMARY:
This study will evaluate post-operative pain in patients undergoing elective caesarean sections based on the method of fascial closure. Patients will be randomised into one of three groups based upon the method of fascial closure and will be followed up over a 10 week period evaluating analgesia use in the acute setting, and also following up with pain scores using a visual analogue score throughout the follow-up period.

DETAILED DESCRIPTION:
Participants will be approached prior to their elective caesarean section to be consented. If they agree to be a part of the study, they will then be randomised into one of three groups based upon the method of fascial closure after delivery of the foetus and closure of the hysterotomy site:

1. Fascia sutured with #1 polysorb braided absorbable suture, with the knot being superficial to the fascia, starting at the left angle of the fascial incision and closed in a continuous fashion. The contralateral angle is grasped with a kocher clamp and the suture is then tied behind the angle ensuring adequate closure.
2. Fascia sutured using #1 polysorb braided absorbable suture with a superficial knot, starting at the left angle and closed in a continuous fashion until the suture is above the right rectus abdominis muscle belly. A second #1 polysorb braided absorbable suture is tied behind the right angle with a superficial knot and run across in a continuous fashion to meet the opposing suture which are then tied together.
3. Fascia sutured using #1 polysorb braided absorbable suture with a buried knot below the fascia starting at the left angle and closed in a continuous fashion until the suture overlies the right rectus abdominis muscle belly. A second #1 polysorb braided absorbable suture is then tied behind the right angle with a buried knot below the fascia and run across in a continuous fashion to meet the opposing suture which are then tied together.

The remainder of the caesarean section is completed in the standard fashion.

Subsequent to this, patients are followed up with a modified brief pain inventory on post-operative day #1, day #7, day #14, day #42 and day #70 to evaluate their pain in the post-operative period. In addition, whilst being inpatients, participant's analgesia use is evaluated using the medication administration record within the unit.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy undergoing elective lower segment caesarean section via a Pfannenstiel incision.
* Caesarean section done via regional anaesthesia (i.e. spinal regional anaesthesia, epidural anaesthesia, combo-spinal+epidural)

Exclusion Criteria:

* Multiple pregnancy
* General anaesthesia
* Caesarean section through laparotomy incision
* History of chronic pain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 450 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score for Pain | Post-operative day #1 and 2, 2, 6, and 10 weeks post-operatively.
  Participants will be asked to fill in a modified MD Anderson Brief Pain Inventory questionnaire with questions related to their overall pain using a visual analogue score ranking from 0 (no pain) to 10 (worst pain imaginable). A higher score will delineate poorer pain control. This questionnaire can be found the attached protocol under "Appendix C". The time points at which these will be measured is on post-operative day #1 and 2, as well as at 2, 6, and 10 weeks post-operatively. We aim to observe a change in the overall pain between groups.
Analgesia use | 48-72 hours
  Will record opioid and non-opioid analgesia use as participants remain in hospital.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT04999670/Prot_SAP_ICF_000.pdf